CLINICAL TRIAL: NCT04574869
Title: A Randomized, Double-Blind, Placebo-Controlled, Two-Part Study to Evaluate the Safety, Tolerability, Preliminary Efficacy, PK, & PD of RLS-0071 in Patients With Acute Lung Injury Due to COVID-19 Pneumonia in Early Respiratory Failure
Brief Title: A Study of RLS-0071 in Patients With Acute Lung Injury Due to COVID-19 Pneumonia in Early Respiratory Failure
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Low probability of enrolling patients prior to expiry of study drug.
Sponsor: ReAlta Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: RLS-0071-102
Record Dates: First submitted 2020-09-16; First posted 2020-10-05 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Acute Lung Injury; ALI; COVID-19
Keywords: Acute Lung Injury; Sars-CoV2; COVID-19; COVID-19 pneumonia; Early Respiratory Failure; ALI
MeSH Terms: conditions — Acute Lung Injury; COVID-19; Respiratory Insufficiency | interventions — RLS-0071

STUDY DESIGN:
Intervention Model Description: Study intervention, RLS-0071 or placebo, will be administered as an IV infusion over 30 minutes (± 10 minutes).
  The following dose groups are planned:
  Part A (Single-Ascending Dose):
  * Cohort 1: low dose (single infusion) vs. placebo
  * Cohort 2: high dose (single infusion) vs. placebo
  Part B (Multiple-Ascending Dose):
  * Cohort 3: low dose administered q8 hours (± 1 hour) vs. placebo for 3 days (9 doses)
  * Cohort 4: high dose administered q8 hours (± 1 hour) vs. placebo for 3 days (9 doses)
Who Masked: Participant, Investigator
Masking Description: This study is a double-blinded and randomized study. Pharmacy staff will mask infusion bags and lines to maintain the study blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental)
  Interventions: Drug: RLS-0071 10 mg/kg; Drug: Placebo
- Cohort 2 (Experimental)
  Interventions: Drug: RLS-0071 40 mg/kg; Drug: Placebo
- Placebo Cohorts 1 and 2 (Placebo Comparator): Placebo will be administered at the same volume and duration of IV infusion corresponding to the cohort dosing schedule.
  Interventions: Drug: Placebo
- Cohort 3 (Experimental)
  Interventions: Drug: Placebo; Drug: RLS-0071 10 mg/kg
- Cohort 4 (Experimental)
  Interventions: Drug: Placebo; Drug: RLS-0071 40 mg/kg
- Placebo Cohorts 3 and 4 (Placebo Comparator): Placebo will be administered at the same volume and duration of IV infusion corresponding to the cohort dosing schedule.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RLS-0071 10 mg/kg — Single dose IV infusion of 10 mg/kg RLS-0071
  Arms: Cohort 1
Drug: RLS-0071 40 mg/kg — Single dose IV infusion of 40 mg/kg RLS-0071
  Arms: Cohort 2
Drug: Placebo — The placebo control will be commercial sterile saline (0.9% Sodium Chloride Injection, United States Pharmacopoeia [USP]).
Drug: RLS-0071 10 mg/kg — Multiple dose IV infusion of 10 mg/kg RLS-0071 administered every 8 hours for approximately 3 days (9 consecutive doses)
  Arms: Cohort 3
Drug: RLS-0071 40 mg/kg — Multiple dose IV infusion of 40 mg/kg RLS-0071 administered every 8 hours for approximately 3 days (9 consecutive doses)
  Arms: Cohort 4

SUMMARY:
The aim of this study will test the safety, tolerability, and efficacy of RLS-0071 for approximately 28 days in comparison to a placebo control in patients with acute lung injury due to COVID-19 pneumonia in early respiratory failure.

Patients will be randomized and double-blinded for two parts, a single-ascending dose (SAD) part and a multiple-ascending dose (MAD) part.

The name of the study drug involved in this study is: RLS-0071.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 based on positive SARS-CoV-2 viral RNA PCR or antigen test.
* Hypoxemia.
* Radiographic evidence of opacification consistent with viral-related pneumonia.
* Weight less than 150 kg.
* Provide written informed consent.

Exclusion Criteria:

* Endotracheal intubation and mechanical ventilation.
* Noninvasive positive pressure ventilation without endotracheal intubation.
* Requires chronic oxygen therapy.
* Treatment with conventional synthetic disease-modifying antirheumatic drugs (DMARDs)/immunosuppressive agents for ≥ 4 weeks duration within 3 months prior to the Screening visit.
* Use of oral corticosteroids in a dose higher than prednisone 15 mg or equivalent per day for ≥ 4 weeks duration within 3 months prior to the Screening visit.
* Systemic autoimmune disease.
* Participation in any clinical research study evaluating an investigational product or therapy within 3 months prior to the Screening visit,
* Presence of any of the following abnormal laboratory values at Screening: absolute neutrophil count < 2,000/mm3, aspartate aminotransferase or alanine aminotransferase > 5 × upper limit of normal (ULN), platelets < 50,000/mm3.
* D-dimer > 2 × ULN at Screening, as evidence of potential disseminated intravascular coagulation (DIC).
* Has confounding medical conditions, including poorly controlled diabetes, uncontrolled New York Heart Association Class III congestive heart failure, clinically significant arrhythmias not controlled by medication, idiopathic pulmonary fibrosis, interstitial lung disease, or chronic obstructive pulmonary disease.
* Has bacterial sepsis currently or suspicion thereof.
* Has cancer currently and is receiving active treatment (including radiation therapy or chemotherapy) or malignancy within the last 5 years, with the exception of curable cancer (eg, basal or squamous cell skin cancer, cervical cancer in situ, nonmedullary thyroid carcinoma) that has been adequately treated (eg, excision).
* Prior history of myocardial infarction or angina, stroke or transient ischemic attack (TIA), pulmonary embolism or deep vein thrombosis.
* Is moribund and not expected to survive 48 hours following Screening or for whom no further aggressive treatment such as mechanical ventilation is planned.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of Adverse Events, including Serious Adverse Events, by treatment group and dose level, including the frequency of premature discontinuation of study intervention due to Adverse Events. | Through study completion at Day 28 following last dose.

SECONDARY OUTCOMES:
Incidence of clinically significant changes from baseline in clinical laboratory values, ADA, autoantibody panel, vital signs, physical examination, ECG, radiography, and concomitant medications. | Through study completion at Day 28 following last dose; (if positive ADA/antibodies, Day 90 and Day 180 following last dose).
Number of patients with positive ADA titers after receiving a single dose (Part A) or multiple doses (Part B) of RLS-0071. | Through study completion at Day 28 following last dose; (if positive ADA/antibodies, Day 90 and Day 180 following last dose).
Estimates of single-dose maximum plasma concentration (Cmax) for RLS-0071. | Pre-Dose (within 30 minutes before start of dosing), 5 and 30 minutes after start of dosing, and 1, 2, 3, 4, 5, 6, 7, 8,12, 18, 24, 36, and 48 hours after the start of dosing, up to 28 days following last dose.
Estimates of single-dose time to maximum plasma concentration (Tmax) for RLS-0071. | Pre-Dose (within 30 minutes before start of dosing), 5 and 30 minutes after start of dosing, and 1, 2, 3, 4, 5, 6, 7, 8,12, 18, 24, 36, and 48 hours after the start of dosing, up to 28 days following last dose.
Estimates of single-dose minimum plasma concentration (Cmin) for RLS-0071. | Pre-Dose (within 30 minutes before start of dosing), 5 and 30 minutes after start of dosing, and 1, 2, 3, 4, 5, 6, 7, 8,12, 18, 24, 36, and 48 hours after the start of dosing, up to 28 days following last dose.
Estimates of single-dose area under the plasma concentration-time curve (AUC) for RLS-0071. | Pre-Dose (within 30 minutes before start of dosing), 5 and 30 minutes after start of dosing, and 1, 2, 3, 4, 5, 6, 7, 8,12, 18, 24, 36, and 48 hours after the start of dosing, up to 28 days following last dose.
Estimates of single-dose apparent total volume of distribution for RLS-0071. | Pre-Dose (within 30 minutes before start of dosing), 5 and 30 minutes after start of dosing, and 1, 2, 3, 4, 5, 6, 7, 8,12, 18, 24, 36, and 48 hours after the start of dosing, up to 28 days following last dose.
Estimates of single-dose apparent total body clearance for RLS-0071. | Pre-Dose (within 30 minutes before start of dosing), 5 and 30 minutes after start of dosing, and 1, 2, 3, 4, 5, 6, 7, 8,12, 18, 24, 36, and 48 hours after the start of dosing, up to 28 days following last dose.
Estimates of single-dose apparent first-order terminal elimination half-life for RLS-0071. | Pre-Dose (within 30 minutes before start of dosing); 30 minutes after the start of dosing; and 1, 2, 4, 6, 12, 18, 24, 36, and 48 hours after the start of dosing. The last PK sample will be taken 48 hours following the last dosing (the 9th infusion
Estimates of multiple-dose maximum plasma concentration (Cmax) for RLS-0071. | Pre-Dose (within 30 minutes before start of dosing); 30 minutes after the start of dosing; and 1, 2, 4, 6, 12, 18, 24, 36, and 48 hours after the start of dosing. The last PK sample will be taken 48 hours following the last dosing (the 9th infusion).
Estimates of multiple-dose peak time to maximum plasma concentration (Tmax) for RLS-0071. | Pre-Dose (within 30 minutes before start of dosing); 30 minutes after the start of dosing; and 1, 2, 4, 6, 12, 18, 24, 36, and 48 hours after the start of dosing. The last PK sample will be taken 48 hours following the last dosing (the 9th infusion).
Estimates of multiple-dose area under the plasma concentration-time curve (AUC) for RLS-0071. | Pre-Dose (within 30 minutes before start of dosing); 30 minutes after the start of dosing; and 1, 2, 4, 6, 12, 18, 24, 36, and 48 hours after the start of dosing. The last PK sample will be taken 48 hours following the last dosing (the 9th infusion).
Estimates of multiple-dose average plasma drug concentration observed (Cavg) for RLS-0071. | Pre-Dose (within 30 minutes before start of dosing); 30 minutes after the start of dosing; and 1, 2, 4, 6, 12, 18, 24, 36, and 48 hours after the start of dosing. The last PK sample will be taken 48 hours following the last dosing (the 9th infusion).
Estimates of multiple-dose trough concentration prior to dose administration (Ctrough). | Pre-Dose (within 30 minutes before start of dosing); 30 minutes after the start of dosing; and 1, 2, 4, 6, 12, 18, 24, 36, and 48 hours after the start of dosing. The last PK sample will be taken 48 hours following the last dosing (the 9th infusion).
Estimates of multiple-dose apparent total volume of distribution for RLS-0071. | Pre-Dose (within 30 minutes before start of dosing); 30 minutes after the start of dosing; and 1, 2, 4, 6, 12, 18, 24, 36, and 48 hours after the start of dosing. The last PK sample will be taken 48 hours following the last dosing (the 9th infusion).
Estimates of multiple-dose apparent first-order terminal elimination half-life for RLS-0071. | Pre-Dose (within 30 minutes before start of dosing); 30 minutes after the start of dosing; and 1, 2, 4, 6, 12, 18, 24, 36, and 48 hours after the start of dosing. The last PK sample will be taken 48 hours following the last dosing (the 9th infusion).
Assessment of dose response relationship of single and multiple doses of RLS-0071 on C1q levels and the complement activity assay. | Through study completion at Day 28 following last dose.
Overall survival. | Through Day 15 and through study completion at Day 28 following last dose.
Incidence of progression to respiratory failure requiring mechanical ventilation. | Days on ventilation while in the hospital through study completion at Day 28.
Incidence of transfer to the ICU. | Through Day 15 following last dose; through study completion at Day 28 following last dose; and duration of ICU stay days in the hospital post-dose through study completion at Day 28.
Duration of hospitalization after treatment (days). | Through study completion at Day 28 following last dose.
Incidence, severity, and duration after treatment (days) of fever (≥ 39.0°C). | Through study completion at Day 28 following last dose.
Incidence, severity, and duration after treatment (days) of cough per investigator assessment of CTCAE's latest version. | Through study completion at Day 28 following last dose.
Duration of requirement for supplemental oxygen after treatment (days). | Through study completion at Day 28 following last dose.
PaO2/FiO2 | Through study completion at Day 28 following last dose.
Incidence, severity, and duration after treatment (days) of new cardiovascular events as assessed by the investigator (e.g. myocardial infarction, stroke, TIA, ischemic limb) with CTCAE's latest version. | Through Day 15 and through study completion at Day 28 following last dose.
Incidence, severity, and duration after treatment (days) of respiratory acidosis as assessed by the investigator with CTCAE's latest version. | Through Day 15 and through study completion at Day 28 following last dose.
Incidence and duration after treatment (days) of dialysis. | Through Day 15 and through study completion at Day 28 following last dose.
  Dialysis will be assessed by the investigator with CTCAE's latest version.
Levels of complement activity (eg, CH50). | Through study completion at Day 28 following last dose.
Levels of C1q (free and bound to RLS-0071). | Through study completion at Day 28 following last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Kenji Cunnion, MD, MPH, Study Chair — ReAlta Life Sciences, Inc.; Linda Dell, Study Director — ReAlta Life Sciences, Inc.
Locations (1):
- Henry Ford Health Systems, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343